CLINICAL TRIAL: NCT07326189
Title: A Prospective, Multicenter, Single-Arm Study on the Efficacy and Safety of Preoperative Right Hepatic Artery Embolization Combined With Surgical Resection for Locally Advanced Bismuth IIIb and IV Perihilar Cholangiocarcinoma
Brief Title: Preoperative Right Hepatic Artery Embolization for Locally Advanced Bismuth IIIb and IV Perihilar Cholangiocarcinoma
Acronym: PHAE-PHCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-989-02
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Cholangiocarcinoma Non-resectable
Keywords: Perihilar cholangiocarcinoma; Hepatic artery embolization; Vascular invasion; Surgical conversion; Radical resection
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preoperative Right Hepatic Artery Embolization + Surgery (Experimental): Participants receive preoperative selective embolization of the tumor-involved right hepatic artery, followed 2-4 weeks later by radical left hepatectomy or left trisectionectomy with resection of the involved artery without reconstruction.
  Interventions: Procedure: Preoperative Right Hepatic Artery Embolization

INTERVENTIONS:
Procedure: Preoperative Right Hepatic Artery Embolization — Participants receive preoperative selective embolization of the tumor-involved right hepatic artery, followed 2-4 weeks later by radical left hepatectomy or left trisectionectomy with resection of the involved artery without reconstruction.

SUMMARY:
This is a prospective, multicenter, single-arm study investigating the efficacy and safety of preoperative right hepatic artery embolization (PHAE) followed by surgical resection in patients with locally advanced Bismuth IIIb or IV perihilar cholangiocarcinoma (PHCC) involving the right hepatic artery. The standard treatment for such cases is often considered unresectable due to the high risk of hepatic ischemia after arterial resection without reconstruction. This study proposes a strategy: preoperative embolization of the tumor-involved right hepatic artery to stimulate the development of collateral arterial circulation (e.g., from the right inferior phrenic artery), enabling subsequent radical resection of the right hepatic artery without reconstruction. The primary objective is to evaluate the 1-year overall survival rate. Secondary objectives include surgical conversion rate, R0 resection rate, 1-year/3-year recurrence-free survival, 3-year overall survival rate and safety assessment. A total of 33 participants will be enrolled across multiple centers in China.

DETAILED DESCRIPTION:
This study aims to validate a novel surgical strategy for locally advanced Bismuth IIIb or IV perihilar cholangiocarcinoma (PHCC) where the tumor involves the right hepatic artery (RHA), rendering the tumor conventionally unresectable due to the high risk of postoperative right hepatic lobe ischemia if the artery is resected without reconstruction. The intervention involves preoperative selective embolization of the tumor-involved RHA using coils. This procedure is intended to induce the development of collateral arterial supply to the right liver lobe from extrahepatic arteries (e.g., right inferior phrenic, adrenal, intercostal arteries) over a 2-4 week period. Following confirmation of collateral circulation via imaging, patients undergo radical left hepatectomy or left trisectionectomy with en-bloc resection of the involved RHA without arterial reconstruction. The study employs a single-arm design. The primary endpoint is the 1-year overall survival (OS) . The study is designed to detect an improvement to 75%, compared to a historical control rate of 54% observed with chemoimmunotherapy for unresectable disease. Secondary endpoints include surgical conversion rate, R0 resection rate, 1-year/3-year recurrence-free survival (RFS), 3-year OS, and safety profiles (incidence of liver abscess, bile leak, post-hepatectomy liver failure, and other Clavien-Dindo ≥ Grade III complications). The study involves multiple phases: screening/preparation (including biliary drainage and portal vein embolization if needed), the PHAE procedure, radical surgery (2-4 weeks post-PHAE), and a 3-year follow-up period. Statistical analysis will be performed on the intention-to-treat (FAS), per-protocol (PPS), and safety (SS) populations.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age 18-80 years.
* Clinical diagnosis of Bismuth IIIb or IV perihilar cholangiocarcinoma, deemed suitable for radical resection via left hepatectomy or left trisectionectomy.
* Imaging (CTA/MRA) confirms tumor invasion of the right hepatic artery (RHA) that is assessed as "unable to be safely reconstructed after resection" (e.g., involvement of RHA branches or requiring vascular graft for reconstruction).
* Portal vein on the side of the future liver remnant is not invaded or is reconstructable.
* ECOG performance status 0-1.
* Child-Pugh score ≤ 7 (Class A or B).
* Adequate organ function (bone marrow, liver, kidney) as per protocol-defined laboratory values.
* Expected survival ≥ 12 weeks.

Exclusion Criteria:

* Evidence of distant metastasis (M1).
* History of other malignancies within the past 5 years (except cured basal cell carcinoma or cervical carcinoma in situ).
* Severe cardiac, pulmonary, renal, or cerebrovascular disease as specified in the protocol (e.g., recent myocardial infarction, severe COPD, chronic renal failure stage ≥ III).
* Uncontrolled active infection or diabetes.
* Pregnancy or lactation.
* Allergy to iodinated contrast media.
* Postoperative pathology confirms non-cholangiocarcinoma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
1-Year Overall Survival | 1 year post-surgery
  The proportion of patients alive at 1 year after the radical surgery date. Overall survival is defined as the time from surgery to death from any cause.

SECONDARY OUTCOMES:
Surgical Conversion Rate | At the time of surgery
  The proportion of enrolled patients who successfully undergo radical resection.
R0 Rate | At the time of surgery
  The proportion of resected patients achieving microscopically negative cut margins at the axial and radial of bile duct tumor.
1-Year and 3-Year Recurrence-Free Survival Rate | 1 year and 3 years post-surgery
  The proportion of patients alive and free of tumor recurrence at 1 and 3 years after surgery. Recurrence-free survival is defined as the time from surgery to the first documented recurrence or death from any cause.
3-Year Overall Survival | 3 years post-surgery
  The proportion of patients alive at 3 years after the radical surgery date.
Incidence of Major Complications (Clavien-Dindo ≥ Grade III) | 90 days post-surgery
  The proportion of patients experiencing post-procedural (embolization or surgery) complications graded as Clavien-Dindo III or higher within 90 days after surgery.

REFERENCES:
- [Background] Mizuno T, Ebata T, Yokoyama Y, Igami T, Yamaguchi J, Onoe S, Watanabe N, Kamei Y, Nagino M. Combined Vascular Resection for Locally Advanced Perihilar Cholangiocarcinoma. Ann Surg. 2022 Feb 1;275(2):382-390. doi: 10.1097/SLA.0000000000004322. PMID 32976284
- [Background] Li B, Li Z, Qiu Z, Qin Y, Gao Q, Ao J, Ma W, Jiang X. Surgical treatment of hilar cholangiocarcinoma: retrospective analysis. BJS Open. 2023 May 5;7(3):zrad024. doi: 10.1093/bjsopen/zrad024. PMID 37194459
- [Background] Kelley RK, Ueno M, Yoo C, Finn RS, Furuse J, Ren Z, Yau T, Klumpen HJ, Chan SL, Ozaka M, Verslype C, Bouattour M, Park JO, Barajas O, Pelzer U, Valle JW, Yu L, Malhotra U, Siegel AB, Edeline J, Vogel A; KEYNOTE-966 Investigators. Pembrolizumab in combination with gemcitabine and cisplatin compared with gemcitabine and cisplatin alone for patients with advanced biliary tract cancer (KEYNOTE-966): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 3;401(10391):1853-1865. doi: 10.1016/S0140-6736(23)00727-4. Epub 2023 Apr 16. PMID 37075781
- [Background] Kang MJ, Jang JY, Chang J, Shin YC, Lee D, Kim HB, Kim SW. Actual Long-Term Survival Outcome of 403 Consecutive Patients with Hilar Cholangiocarcinoma. World J Surg. 2016 Oct;40(10):2451-9. doi: 10.1007/s00268-016-3551-9. PMID 27206402
- [Background] Burris HA 3rd, Okusaka T, Vogel A, Lee MA, Takahashi H, Breder V, Blanc JF, Li J, Bachini M, Zotkiewicz M, Abraham J, Patel N, Wang J, Ali M, Rokutanda N, Cohen G, Oh DY. Durvalumab plus gemcitabine and cisplatin in advanced biliary tract cancer (TOPAZ-1): patient-reported outcomes from a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2024 May;25(5):626-635. doi: 10.1016/S1470-2045(24)00082-2. PMID 38697156
- [Background] Benson AB 3rd, D'Angelica MI, Abrams T, Ahmed A, Akce M, Anaya DA, Anders R, Are C, Aye L, Bachini M, Baker M, Binder D, Brown DB, Burgoyne A, Castellanos J, Cloyd J, Cullinan D, Franses J, Glazer ES, Harris W, Iyer R, Jennings L, Kelley RK, Khan S, Levine M, Melstrom L, Palta M, Raman S, Ronnekleiv-Kelly S, Sahai V, Stein S, Stephans K, Thanikachalam K, Turk A, Vauthey JN, Venook AP, Yano M, Yopp A, Zhao K, Schonfeld R, Hochstetler C. Biliary Tract Cancers, Version 2.2025, NCCN Clinical Practice Guidelines In Oncology. J Natl Compr Canc Netw. 2025 Sep;23(9):403-418. doi: 10.6004/jnccn.2025.0042. PMID 40930144